CLINICAL TRIAL: NCT07331610
Title: Effects Of Down-Dog Yoga On Pain And Posture In Children With Nonspecific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUHAMMAD HAROON UR RAHMAN
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
Keywords: PaediatricYoga,DownwardDog Pose,Postural Assessment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Down dog yoga with routine physical therapy group (Experimental): Warm-Up Complementary Yoga Poses
  Other supportive poses will be integrated to enhance the effects of Down-Dog Yoga:
  Child's Pose Cool Down and Relaxation
  Interventions: Other: down dog yoga
- Routine physical therapy group (Active Comparator): The control group will receive standard conventional physiotherapy designed for the management of nonspecific low back pain in children. This intervention focuses on general stretching, strengthening, and postural correction exercises that are commonly used in clinical pediatric rehabilitation Warm-Up Bird-dog Gentle stretching: Focus on back, hips, and hamstrings Deep breathing and relaxation: In seated or lying down position
  Interventions: Other: down dog yoga

INTERVENTIONS:
Other: down dog yoga — experimenbtal group was given down dog yoga protocol along with back and trunk isometric and trunk streching control group wasa givcen standard phyiotherapy intervention total 2 session will given each week consisting of 30 mints
  Other Names: No intervention

SUMMARY:
To manage back pain and correct postural imbalances in children, Downward-Facing Dog (Adho Mukha Svanasana) promotes flexibility, core strength, and spinal alignment.

Traditional physiotherapy may seem repetitive and less engaging for kids. Yoga offers a developmentally appropriate, non-invasive, and enjoyable alternative. Studying its effectiveness could provide a simple, affordable, and accessible therapy option.

DETAILED DESCRIPTION:
School-aged children are increasingly experiencing nonspecific low back pain (NSLBP) as a result of sedentary lifestyles, bad posture, and inactivity. This illness frequently results in discomfort, decreased engagement in physical activities, and a lower standard of living. Preventing chronic pain and long-term incapacity requires early intervention.

The benefits of yoga as a physical and mental treatment for musculoskeletal issues are becoming more widely acknowledged. A basic yoga stance that develops the core muscles, improves spinal alignment, and extends the body's posterior chain is the Down-Dog pose. Research on its use in the paediatric population is few, despite the fact that its advantages in adults are widely established. The purpose of this study is to investigate how well Down-Dog yoga helps children with NSLBP with their pain management and posture. Participants in this randomized controlled experiment will be school-age children (8-14 years old) with a clinical diagnosis of nonspecific low back pain. A control group will get traditional stretching and posture correction activities, while an experimental group will practice Down-Dog yoga. Participants will be randomly assigned to either group.

During a six-week period, both interventions will be given three times a week for 30 minutes each. The Plumb Line Test and Modified Schober's Test will be used to assess postural alignment, and the Visual Analog Scale (VAS) will be used to gauge pain levels.

Children's everyday functioning will be evaluated as a result of the intervention using the Paediatric Quality of Life Inventory (PedsQL). Data will be gathered both before and after the intervention, and the proper statistical methods will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

Children aged 8 to 14 years Actively enrolled in a regular school setting. Clinical diagnosis of non-specific low back pain Pain duration of at least 4 weeks but less than 6 months. Self-reported pain of ≥3 on a 10-point Visual Analog Scale or age-appropriate pain scale Presence of observable postural misalignment

Exclusion Criteria:

History or evidence of spinal deformity Structural abnormalities History of neuromuscular disorders, cerebral palsy, or epilepsy Trauma, fractures, or surgery to the spine or lower limbs in the last 6 months.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
plumb line for posture correction | Baseline and after 6 weeks
  the individual stands upright next to a vertical plumb line (or against a grid or wall) so that their posture can be visually evaluated. Key anatomical landmarks such as the ear lobe, shoulder, hip, knee, and ankle are observed in relation to the plumb line to detect deviations from normal alignment. It is a non-invasive, quick, and cost-effective method commonly used in physiotherapy and rehabilitation settings to identify postural imbalances.

CONTACTS AND LOCATIONS:
Overall Officials: muhammad haroon, dpt, Principal Investigator — Riphah International University, Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: oga may be a beneficial form of exercise in the school-based setting for improving balance and flexibility in healthy children. — https://pubmed.ncbi.nlm.nih.gov/31733751/